CLINICAL TRIAL: NCT04539002
Title: Aerobic Exercise to Improve Mobility in Multiple Sclerosis: Optimizing Design and Execution for a Full-scale Multimodal Remyelination Clinical Trial
Brief Title: Aerobic Exercise for Remyelination in Multiple Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Portland VA Medical Center (U.S. Federal Agency); Oregon Clinical and Translational Research Institute (Other); Myelin Repair Foundation (Unknown); EMD Serono (Industry); Medical Research Foundation, Oregon (Other)
Responsible Party: Principal Investigator, Lindsey Wooliscroft, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00021045; K23HD101667 (NIH); UL1TR002369 (NIH)
Record Dates: First submitted 2020-08-26; First posted 2020-09-04 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis; Sclerosis; Demyelinating Diseases; Autoimmune Diseases of the Nervous System; Nervous System Diseases; Demyelinating Autoimmune Diseases, CNS; Exercise
Keywords: Exercise; Aerobic Exercise; Remyelination; Neural Repair; Mobility
MeSH Terms: conditions — Multiple Sclerosis; Sclerosis; Demyelinating Diseases; Autoimmune Diseases of the Nervous System; Nervous System Diseases; Demyelinating Autoimmune Diseases, CNS; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The first 44 participants with spinal cord injury related to multiple sclerosis (MS) will be randomized in a 1:1 ratio to a 24-week aerobic exercise intervention on a stationary ergometer or an MS education control group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Single-blind, randomized, controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MS: Cycle (Experimental): Twenty-two participants in the clinical trial arm will be randomized to MS:Cycle: an aerobic exercise intervention on a stationary ergometer. Participants will exercise thrice weekly for 30 minutes with graded supervision for 24 weeks.
  Interventions: Behavioral: Aerobic exercise
- MS: Take Control (Active Comparator): Twenty-two participants in the clinical trial arm will be randomized to MS: Take Control (MSTC): a monthly, hour-long MS education control group led by a trained facilitator.
  Interventions: Behavioral: Education Group Control

INTERVENTIONS:
Behavioral: Aerobic exercise — Aerobic exercise performed on a stationary ergometer for 30 minutes, thrice weekly, with graded supervision. Participants will participate in the intervention over 24 weeks.
  Arms: MS: Cycle
Behavioral: Education Group Control — A monthly, hour-long, class over various MS topics and symptoms, led by a trained facilitator.
  Arms: MS: Take Control

SUMMARY:
This is a clinical trial to determine the feasibility of a stationary aerobic cycling intervention and explore if aerobic exercise independently promotes remyelination in people with multiple sclerosis (MS).

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is the most common non-traumatic disabling neurologic condition of young adulthood, affecting more than 2.5 million people worldwide. Permanent disability in MS is caused by recurrent demyelination due to episodic inflammation, followed by neuronal damage, axonal degeneration, and progressive failure of remyelination. There is an urgent need to restore activity and participation in people with MS (pwMS), and remyelination is the most promising therapeutic strategy to accomplish this goal.

Remyelination in pwMS will likely require integration of pharmacologic and rehabilitative approaches to ensure effective remyelination of appropriate neural pathways. Aerobic exercise is an ideal complement to remyelinating medications because aerobic exercise 1) improves walking function in pwMS, and 2) promotes remyelination in animal models both independently and synergistically with medications. However, there are many unknowns that need to be addressed before aerobic exercise can be explored in multimodal clinical trials for remyelination. First, it is imperative to understand how myelination impacts disability in MS, as many other factors could contribute to reduced activity and participation. Additionally, as remyelination occurs over 12 to 24 weeks, it is imperative to establish the feasibility of similar duration of aerobic exercise interventions, and explore if exercise independently influences established remyelination outcomes before integration into multimodal strategies.

This is a randomized, single-blind, parallel clinical trial of a 24-week aerobic stationary cycling intervention to determine feasibility and explore if aerobic exercise independently promotes remyelination in pwMS.

ELIGIBILITY:
Inclusion Criteria:

* Physician-confirmed diagnosis of MS based on the 2017 McDonald criteria
* 18-64 years old
* Have access to the internet and a device that can access virtual visits
* (Inclusion criteria to advance to clinical trial) Somatosensory evoked potential (SSEP) latency z-score ≥2 for P40 or inter-side difference in z-score ≥2 for P40

Exclusion Criteria:

* Medical or biophysical conditions that prohibit the use of a cycle ergometer or treadmill (medical readiness to be assessed by the Activity Readiness Questionnaire (PAR-Q)) or achievement of target heart rate.
* Engages in >30 minutes/week of aerobic activity regularly.
* Clinically confirmed MS relapse in the last 3 months.
* Changes in disease modifying therapy (DMT) for MS in the last 6 months.
* Pregnant women.
* Treatment with steroids for MS in the last 30 days.
* Concurrent use of 4-aminopyridine or dalfampridine (medications which can alter SSEP) and unwilling to discontinue it for 2 days prior to SSEP testing.
* Have a known history of severe spinal canal stenosis

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Somatosensory Evoked Potentials (SSEPs) | From baseline to week 24
  Measure of functional myelination of the somatosensory tracts of the spinal cord

SECONDARY OUTCOMES:
6-Minute Timed Walk (6MTW) | From baseline to week 24
  An assessment of exercise tolerance
Timed Up and Go (TUG) | From baseline to week 24
  A test of walking agility
Timed 25-Foot Walk (T25FW) | From baseline to week 24
  A test of walking speed
Fall frequency | From baseline to week 24
  A self-report of fall frequency over the last 30 days
9 Hole Peg Test | From baseline to week 24
  A test of upper extremity and arm function
Multiple Sclerosis Functional Composite (MSFC) | From baseline to week 24
  Composite measure of walking speed, upper extremity function and cognition.
Virtual aerobic exercise intervention adherence | From baseline to week 24
  Defined as participation in at least 80% of the exercise sessions in the trial
Virtual education control group adherence | From baseline to week 24
  Defined as participation in at least 80% of the education group sessions in the trial
Average heart rate (HR) zone during exercise sessions | From baseline to week 24
  Average HR zone during exercise sessions
Brain Myelin Water Fraction (MWF) | From baseline to week 24
  MWF imaging of the corpus callosum, internal capsules and MS lesions
Symbol Digit Modalities Test (SDMT) | From baseline to week 24
  A test of cognitive function
VO2 max | From baseline to week 24
  A test of aerobic fitness
7-site skinfold test | From baseline to week 24
  A test of body composition
Modified Fatigue Impact Scale (MFIS) | From baseline to week 24
  A patient reported outcome of fatigue severity with a range of 0-84 (higher scores indicate more fatigue).
Pain Effects Scale (PES) | From baseline to week 24
  A patient reported outcome of pain with a range of 6-30 (higher scores indicate a greater impact of pain on a person's mood or behavior).
Health-related quality of life (QoL) | From baseline to weeks 24
  Neuro-QoL questionnaires of upper and lower extremity function, depression, sleep, and self efficacy
International Physical Activity Questionnaire Short Form (IPAQ-SF) | From baseline to week 24
  A patient reported outcome of physical activity

OTHER OUTCOMES:
Patient Determined Disease Steps (PDDS) | Baseline
  A patient reported outcome of MS disability ranging from 0-8 (with higher scores indicating increased disability).
Activity Readiness Questionnaire (PAR-Q) | Baseline and 12 weeks
  An assessment of safety to participate in exercise
6-Minute Timed Walk (6MTW) | From baseline to week 12
  An assessment of exercise tolerance
Timed Up and Go (TUG) | From baseline to week 12
  A test of walking agility
Timed 25-Foot Walk (T25FW) | From baseline to week 12
  A test of walking speed
Fall frequency | From baseline to week 12
  A self-report of fall frequency over the last 30 days
9 Hole Peg Test | From baseline to week 12
  A test of upper extremity and arm function
Multiple Sclerosis Functional Composite (MSFC) | From baseline to week 12
  Composite measure of walking speed, upper extremity function and cognition.
Symbol Digit Modalities Test (SDMT) | From baseline to week 12
  A test of cognitive function
Modified Fatigue Impact Scale (MFIS) | From baseline to week 12
  A patient reported outcome of fatigue severity with a range of 0-84 (higher scores indicate more fatigue).
Pain Effects Scale (PES) | From baseline to week 12
  A patient reported outcome of pain with a range of 6-30 (higher scores indicate a greater impact of pain on a person's mood or behavior).
Somatosensory Evoked Potentials (SSEPs) | From baseline to week 12
  Measure of functional myelination of the somatosensory tracts of the spinal cord
Strength testing | From baseline to week 24
  Strength of the quadriceps, hamstrings, and hand grip is measured with dynamometers
Strength testing | From baseline to week 12
  Strength of the quadriceps, hamstrings, and hand grip is measured with dynamometers
Health-related quality of life (QoL) | From baseline to weeks 12
  Neuro-QoL questionnaires of upper and lower extremity function, depression, sleep, and self efficacy
International Physical Activity Questionnaire Short Form (IPAQ-SF) | From baseline to week 12
  A patient reported outcome of physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey B Wooliscroft, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wooliscroft L, McCoy S, Hildebrand A, Rooney W, Oken BS, Spain RI, Kuehl KS, Bourdette D, Cameron M. Protocol for an exploratory, randomised, single-blind clinical trial of aerobic exercise to promote remyelination in multiple sclerosis. BMJ Open. 2023 Jan 3;13(1):e061539. doi: 10.1136/bmjopen-2022-061539. PMID 36596632